CLINICAL TRIAL: NCT02844010
Title: Prospective Study to Quantify the Change in Weight at a Pneumonia
Acronym: PneumoniePoids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC14.323
Record Dates: First submitted 2016-07-11; First posted 2016-07-26 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Hospitalisation for Pneumonia
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Weight is written down.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with pneumonia
  Interventions: Other: weighing

INTERVENTIONS:
Other: weighing

SUMMARY:
This study is based on the change in weight of hospitalized patients knowing that the diagnosis of malnutrition based on the presence of at least one clinical or laboratory test which anthropometric measures (Evaluation of diagnostic protein energy malnutrition in hospitalized adults ANAES , Guidelines Department, September 2003; HAS Strategy supported in cases of wasting energy and protein in the elderly April 2007).

The goal of this study is to find the correlation between hospitalization and weight loss, significant risk factors for malnutrition in a situation of community-acquired pneumonia infection.

ELIGIBILITY:
Inclusion Criteria:

* cough
* Fever > 38.5 ° C
* Tachycardia > 100 / Min
* Chest pain lateralized
* Absence of infection high respiratory tract
* Global Impression of Severity
* Fireplace auscultatory signs (rattle crackling)

Exclusion Criteria:

* Pregnant women
* Dialysis patients
* Any patient with home oxygen or under a home care for BPCO stage 3 or 4
* Patients transferred from intensive care
* Patients with severe sepsis and requiring a "filler"
* Enteral or parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Weight history | Few minutes
  The weight of the patient, and weight's history.
Standard biology | Few hours
  C-reactive protein, Albumine, Transthyretin, Oxygen
Severity of pneumonia | Few minutes
  Fine's score or CURB 65
The functional status | Few minutes
  ADL score ; activities daily living

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arnone D, Cavanagh J, Gerber D, Lawrie SM, Ebmeier KP, McIntosh AM. Magnetic resonance imaging studies in bipolar disorder and schizophrenia: meta-analysis. Br J Psychiatry. 2009 Sep;195(3):194-201. doi: 10.1192/bjp.bp.108.059717. PMID 19721106
- [Background] Bamford S, Ward R. Predispositions to approach and avoid are contextually sensitive and goal dependent. Emotion. 2008 Apr;8(2):174-83. doi: 10.1037/1528-3542.8.2.174. PMID 18410191
- [Background] Bradley MM, Sabatinelli D, Lang PJ, Fitzsimmons JR, King W, Desai P. Activation of the visual cortex in motivated attention. Behav Neurosci. 2003 Apr;117(2):369-80. doi: 10.1037/0735-7044.117.2.369. PMID 12708533
- [Background] Bradley MM. Natural selective attention: orienting and emotion. Psychophysiology. 2009 Jan;46(1):1-11. doi: 10.1111/j.1469-8986.2008.00702.x. Epub 2008 Sep 5. PMID 18778317
- [Background] Briggs KE, Martin FH. Target processing is facilitated by motivationally relevant cues. Biol Psychol. 2008 Apr;78(1):29-42. doi: 10.1016/j.biopsycho.2007.12.007. Epub 2008 Jan 4. PMID 18262710
- [Background] Bulot V, Thomas P, Delevoye-Turrell Y. A pre-reflective indicator of an impaired sense of agency in patients with Schizophrenia. Exp Brain Res. 2007 Oct;183(1):115-26. doi: 10.1007/s00221-007-1027-8. Epub 2007 Jul 10. PMID 17619866
- [Background] Cirillo MA, Seidman LJ. Verbal declarative memory dysfunction in schizophrenia: from clinical assessment to genetics and brain mechanisms. Neuropsychol Rev. 2003 Jun;13(2):43-77. doi: 10.1023/a:1023870821631. PMID 12887039
- [Background] Delplanque S, Lavoie ME, Hot P, Silvert L, Sequeira H. Modulation of cognitive processing by emotional valence studied through event-related potentials in humans. Neurosci Lett. 2004 Feb 6;356(1):1-4. doi: 10.1016/j.neulet.2003.10.014. PMID 14746887
- [Background] Ellison-Wright I, Glahn DC, Laird AR, Thelen SM, Bullmore E. The anatomy of first-episode and chronic schizophrenia: an anatomical likelihood estimation meta-analysis. Am J Psychiatry. 2008 Aug;165(8):1015-23. doi: 10.1176/appi.ajp.2008.07101562. Epub 2008 Apr 1. PMID 18381902
- [Background] Goldman-Rakic PS. Working memory dysfunction in schizophrenia. J Neuropsychiatry Clin Neurosci. 1994 Fall;6(4):348-57. doi: 10.1176/jnp.6.4.348. PMID 7841806
- [Background] Frijda, N.H. (1986). The emotions. Cambridge et New-York: Cambridge University Press.
- [Background] Frijda, N.H. (1987). Emotions, cognitive structure, and action tendency. Cognition and Emotion, 1, 115-143.
- [Background] Glahn DC, Laird AR, Ellison-Wright I, Thelen SM, Robinson JL, Lancaster JL, Bullmore E, Fox PT. Meta-analysis of gray matter anomalies in schizophrenia: application of anatomic likelihood estimation and network analysis. Biol Psychiatry. 2008 Nov 1;64(9):774-81. doi: 10.1016/j.biopsych.2008.03.031. Epub 2008 May 16. PMID 18486104
- [Background] Hajcak G, Dunning JP, Foti D. Motivated and controlled attention to emotion: time-course of the late positive potential. Clin Neurophysiol. 2009 Mar;120(3):505-10. doi: 10.1016/j.clinph.2008.11.028. Epub 2009 Jan 20. PMID 19157974
- [Background] Hajcak G, Moser JS, Simons RF. Attending to affect: appraisal strategies modulate the electrocortical response to arousing pictures. Emotion. 2006 Aug;6(3):517-22. doi: 10.1037/1528-3542.6.3.517. PMID 16938092
- [Background] Hajcak G, Molnar C, George MS, Bolger K, Koola J, Nahas Z. Emotion facilitates action: a transcranial magnetic stimulation study of motor cortex excitability during picture viewing. Psychophysiology. 2007 Jan;44(1):91-7. doi: 10.1111/j.1469-8986.2006.00487.x. PMID 17241144
- [Background] Harmon-Jones E, Lueck L, Fearn M, Harmon-Jones C. The effect of personal relevance and approach-related action expectation on relative left frontal cortical activity. Psychol Sci. 2006 May;17(5):434-40. doi: 10.1111/j.1467-9280.2006.01724.x. PMID 16683932
- [Background] Honea R, Crow TJ, Passingham D, Mackay CE. Regional deficits in brain volume in schizophrenia: a meta-analysis of voxel-based morphometry studies. Am J Psychiatry. 2005 Dec;162(12):2233-45. doi: 10.1176/appi.ajp.162.12.2233. PMID 16330585
- [Background] Ha TH, Youn T, Ha KS, Rho KS, Lee JM, Kim IY, Kim SI, Kwon JS. Gray matter abnormalities in paranoid schizophrenia and their clinical correlations. Psychiatry Res. 2004 Dec 30;132(3):251-60. doi: 10.1016/j.pscychresns.2004.05.001. PMID 15664796
- [Background] Ito TA, Larsen JT, Smith NK, Cacioppo JT. Negative information weighs more heavily on the brain: the negativity bias in evaluative categorizations. J Pers Soc Psychol. 1998 Oct;75(4):887-900. doi: 10.1037//0022-3514.75.4.887. PMID 9825526
- [Background] Kasanin J. The acute schizoaffective psychoses. 1933. Am J Psychiatry. 1994 Jun;151(6 Suppl):144-54. doi: 10.1176/ajp.151.6.144. No abstract available. PMID 8192190
- [Background] Maier W, Zobel A, Wagner M. Schizophrenia and bipolar disorder: differences and overlaps. Curr Opin Psychiatry. 2006 Mar;19(2):165-70. doi: 10.1097/01.yco.0000214342.52249.82. PMID 16612197
- [Background] McDonald C, Bullmore E, Sham P, Chitnis X, Suckling J, MacCabe J, Walshe M, Murray RM. Regional volume deviations of brain structure in schizophrenia and psychotic bipolar disorder: computational morphometry study. Br J Psychiatry. 2005 May;186:369-77. doi: 10.1192/bjp.186.5.369. PMID 15863740
- [Background] Ochsner KN, Gross JJ. The cognitive control of emotion. Trends Cogn Sci. 2005 May;9(5):242-9. doi: 10.1016/j.tics.2005.03.010. PMID 15866151
- [Background] Peterson CK, Shackman AJ, Harmon-Jones E. The role of asymmetrical frontal cortical activity in aggression. Psychophysiology. 2008 Jan;45(1):86-92. doi: 10.1111/j.1469-8986.2007.00597.x. Epub 2007 Sep 10. PMID 17850239
- [Background] Phan KL, Taylor SF, Welsh RC, Decker LR, Noll DC, Nichols TE, Britton JC, Liberzon I. Activation of the medial prefrontal cortex and extended amygdala by individual ratings of emotional arousal: a fMRI study. Biol Psychiatry. 2003 Feb 1;53(3):211-5. doi: 10.1016/s0006-3223(02)01485-3. PMID 12559653
- [Background] Phillips ML, Drevets WC, Rauch SL, Lane R. Neurobiology of emotion perception I: The neural basis of normal emotion perception. Biol Psychiatry. 2003 Sep 1;54(5):504-14. doi: 10.1016/s0006-3223(03)00168-9. PMID 12946879
- [Background] Phillips ML, Ladouceur CD, Drevets WC. A neural model of voluntary and automatic emotion regulation: implications for understanding the pathophysiology and neurodevelopment of bipolar disorder. Mol Psychiatry. 2008 Sep;13(9):829, 833-57. doi: 10.1038/mp.2008.65. Epub 2008 Jun 24. PMID 18574483
- [Background] Rich BA, Schmajuk M, Perez-Edgar KE, Pine DS, Fox NA, Leibenluft E. The impact of reward, punishment, and frustration on attention in pediatric bipolar disorder. Biol Psychiatry. 2005 Oct 1;58(7):532-9. doi: 10.1016/j.biopsych.2005.01.006. Epub 2005 Jun 13. PMID 15953589
- [Background] Sander D. et Scherer K.R. (2009). Traité de psychologie des émotions. Dunod édition.
- [Background] Savitz J, Drevets WC. Bipolar and major depressive disorder: neuroimaging the developmental-degenerative divide. Neurosci Biobehav Rev. 2009 May;33(5):699-771. doi: 10.1016/j.neubiorev.2009.01.004. Epub 2009 Jan 21. PMID 19428491
- [Background] Scherer, K.R. (2001). " Appraisal considered as a process of multilevel sequential checking ". In K.R. Scherer, A. Schorr, T. Johm-Stone (éd.), Appraisal Processes in Emotion: Theory, Methods, Research. New York: Oxforf University Press.
- [Background] Schiff BB, Guirguis M, Kenwood C, Herman CP. Asymmetrical hemispheric activation and behavioral persistence: effects of unilateral muscle contractions. Neuropsychology. 1998 Oct;12(4):526-32. doi: 10.1037//0894-4105.12.4.526. PMID 9805322
- [Background] Shenton ME, Dickey CC, Frumin M, McCarley RW. A review of MRI findings in schizophrenia. Schizophr Res. 2001 Apr 15;49(1-2):1-52. doi: 10.1016/s0920-9964(01)00163-3. PMID 11343862
- [Background] Taylor JG. A neural model of the loss of self in schizophrenia. Schizophr Bull. 2011 Nov;37(6):1229-47. doi: 10.1093/schbul/sbq033. Epub 2010 Apr 23. PMID 20418446
- [Background] Vita A, De Peri L, Silenzi C, Dieci M. Brain morphology in first-episode schizophrenia: a meta-analysis of quantitative magnetic resonance imaging studies. Schizophr Res. 2006 Feb 15;82(1):75-88. doi: 10.1016/j.schres.2005.11.004. Epub 2005 Dec 27. PMID 16377156
- [Background] Vuilleumier P, Armony JL, Driver J, Dolan RJ. Distinct spatial frequency sensitivities for processing faces and emotional expressions. Nat Neurosci. 2003 Jun;6(6):624-31. doi: 10.1038/nn1057. PMID 12740580
- [Background] Wright IC, Rabe-Hesketh S, Woodruff PW, David AS, Murray RM, Bullmore ET. Meta-analysis of regional brain volumes in schizophrenia. Am J Psychiatry. 2000 Jan;157(1):16-25. doi: 10.1176/ajp.157.1.16. PMID 10618008